CLINICAL TRIAL: NCT00931151
Title: Effects of Dietary Protein on Undesirable Postprandial Events in Overweight Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement (Other)
Collaborators: National Research Agency, France (Other)
Responsible Party: Principal Investigator, Robert Benamouzig, Professor, Institut National de Recherche pour l'Agriculture, l'Alimentation et l'Environnement
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SURPROL 2
Record Dates: First submitted 2009-07-01; First posted 2009-07-02 (Estimated); Last update posted 2011-08-23 (Estimated); Status verified 2010-03

CONDITIONS: Overweight
MeSH Terms: conditions — Overweight

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Casein (Experimental): Protein source in the high fat meal is casein
  Interventions: Dietary Supplement: Postprandial metabolic and functional measures
- Milk soluble protein (Experimental): Protein source in the high fat meal are milk soluble protein
  Interventions: Dietary Supplement: Postprandial metabolic and functional measures
- Alpha lactalbumin (Experimental): Protein source in the high fat meal is alpha-lactalbumin
  Interventions: Dietary Supplement: Postprandial metabolic and functional measures

INTERVENTIONS:
Dietary Supplement: Postprandial metabolic and functional measures — After ingestion of a high fat meal containing the different protein sources, the subjects undergo a series of measures of endothelial dysfunction and blood and urine sampling for the assessment of proinflammatory cytokines levels and metabolomics determinations.

SUMMARY:
Dietary protein differing by their amino acid composition could modulate undesirable metabolic and functional responses to a meal rich in saturated fat and sugars. This study aims at examining the specific effects of dairy protein with different cysteine contents on the postprandial undesirables effects elicited by the ingestion of a high fat meal in overweight subjects.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 25 and 30
* Waist circumference > 94 cm

Exclusion Criteria:

* Allergy to milk protein
* Abusive drug consumption
* Smoking
* Hypertension, diabetes
* High level of physical activity

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-04; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Endothelial dysfunction | 0-2-4-6 hours (after meal ingestion)

SECONDARY OUTCOMES:
Postprandial inflammation | 0-0.5-1-1.5-2-3-4-6 hours (after meal ingestion)

CONTACTS AND LOCATIONS:
Overall Officials: Robert Benamouzig, MD, Ph. D, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Centre de recherche sur volontaires, Bobigny, France

REFERENCES:
- [Derived] Pujos-Guillot E, Brandolini-Bunlon M, Fouillet H, Joly C, Martin JF, Huneau JF, Dardevet D, Mariotti F. Metabolomics Reveals that the Type of Protein in a High-Fat Meal Modulates Postprandial Mitochondrial Overload and Incomplete Substrate Oxidation in Healthy Overweight Men. J Nutr. 2018 Jun 1;148(6):876-884. doi: 10.1093/jn/nxy049. PMID 29878266
- [Derived] Mariotti F, Valette M, Lopez C, Fouillet H, Famelart MH, Mathe V, Airinei G, Benamouzig R, Gaudichon C, Tome D, Tsikas D, Huneau JF. Casein Compared with Whey Proteins Affects the Organization of Dietary Fat during Digestion and Attenuates the Postprandial Triglyceride Response to a Mixed High-Fat Meal in Healthy, Overweight Men. J Nutr. 2015 Dec;145(12):2657-64. doi: 10.3945/jn.115.216812. Epub 2015 Oct 21. PMID 26491119